CLINICAL TRIAL: NCT05951803
Title: Effectiveness of the Brief Behavioral Intervention for Insomnia in the Teleconsultation Modality (ICBI-TC) on the Symptoms of Anxiety, Depression, Sleep Quality and Quality of Life in Insomniac Patients.
Brief Title: Effectiveness of a Psychological Intervention on Mental Health and Sleep.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Horacio Balam ALvarez Garcia, investigator, Hospital General de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGMexico
Record Dates: First submitted 2023-06-22; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Insomnia Chronic; Anxiety; Depression; Sleep Quality; Life Quality
Keywords: INSOMNIA; ANXIETY; LIFE QUALITY; teleconsultation; LONG COVID
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of equivalence with two groups in parallel (1:1) with repeated measures in pretreatment, posttreatment and follow-up at 3 months
Masking Description: in data analysis, an external investigator will be asked to perform randomization and data processing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Behavioral Intervention in Insomnia through Tele-Consultation (BBII-TC) (Other): Brief therapy organized into four sessions, lasting 60 minutes each, where behavioral therapy techniques are taught (stimulus control, sleep restriction, progressive muscle relaxation, sleep hygiene). The teleconsultation modality is given through the ZOOM platform synchronously.
  Interventions: Behavioral: Brief Behavioral Intervention in Insomnia

INTERVENTIONS:
Behavioral: Brief Behavioral Intervention in Insomnia — Weekly intervention of 4 sessions where behavior therapy techniques are administered, such as stimulus control, sleep hygiene, sleep restriction and progressive muscle relaxation. Each session lasts 60 minutes.
  Other Names: Brief Cognitive Behavioral Therapy for Insomnia

SUMMARY:
Background: The COVID-19 pandemic represented a global public health problem that brought considerable consequences to the physical and mental health of the entire population. Objective: To compare the effectiveness of the brief behavioral intervention for insomnia by teleconsultation (BBII-TC) with the brief behavioral intervention for face-to-face insomnia (BBII) on symptoms of insomnia, anxiety, depression, quality of sleep and life in a sample. of patients with long COVID. Methodology: Randomized controlled trial of equivalence with two groups in parallel (1:1) with repeated measures in pretreatment, posttreatment and follow-up at 3 months. The sample will be composed of male or female participants, in an age range of 18 to 40 years. The sample size was calculated, obtaining a total of 52 participants, the expected effect size is .40, with a significance of 0.05 and a probability error of 80%. Participants in the two groups will be assessed with the following instruments: Sleep Diary, Patient Health Questionnaire 9, Pittsburgh Sleep Quality Index , Insomnia Severity Index, SF-36 Health Survey and Generalized Anxiety Disorder 7; at the beginning and end of treatment; and in a follow-up at 3 months. TData analysis: The Kolmogrov-Smirnov test will be carried out to determine the normality of the data, in case the distribution is parametric, an ANOVA of repeated measures will be carried out for the comparison of data between the pre, post and monitoring for each of the groups; in the event that the data does not have a normal distribution, the Friedman test will be performed for the comparison of repeated measures. Finally, to avoid bias in the data analysis, an external investigator will be asked to perform the randomization and data processing.

DETAILED DESCRIPTION:
Once the sample is composed, the participants will be randomized in a simple computerized way to one of the two groups. A structured clinical interview will be carried out, then they will be given the sleep diary and the instruments will be applied to measure the degree of symptoms of sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Have a personal pathological history of diagnosis of COVID-19 (mild or severe) by PCR test or antigen test in the last 6 months.
* Present symptoms of insomnia.
* Present anxiety symptoms.
* Present symptoms of depression.
* Be between 18 and 40 years old.
* Have digital devices such as a computer, tablet or smartphone with internet access.

Exclusion Criteria:

* Being in psychological or pharmacological treatment to control insomnia, anxiety, depression, at the time of the study.
* Presenting symptoms of another sleep disorder such as obstructive sleep apnea, restless legs syndrome, or sleep disorder due to work hours (1).
* Suffering from cardiorespiratory or neurological sequelae of COVID-19 do not allow the participant to take the treatment.
* Consume psychoactive substances of abuse (Cannabis, cocaine, solvents, cannabidiol).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Sleep diary | 1 week after starting treatment.
  Self-registration format subjectively evaluates the number of sleepless nights, subjective sleep quality, number of awakenings per night, sleep onset latency, and sleep efficacy
Patient Health Questionnaire 9 (PHQ-9) | 1 week after starting treatment.
  Self-applied questionnaire that assesses the presence and severity of depressive symptoms. It is made up of 9 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range of 0 to 27. These scores are interpreted from 0 to 5 (mild), 6 to 10 (moderate), 11 to 15 (moderately severe) and 16 to 27. (severe). Within its psychometric properties, the original version has a high internal consistency with a Cronbach's alpha of 0.86, while the Mexican version was 0.89.
Pittsburgh Sleep Quality Index (PSQI) | 1 week after starting treatment.
  Self-administered questionnaire that assesses sleep quality. It is made up of 24 reagents; the total score has a range of 0 to 21 points; where a total score less than 5 points indicates good sleep quality and a score greater than 5 points is interpreted as poor sleep quality. In the Mexican population, he obtained a Cronbach's Alpha of 0.78.
Insomnia Severity Index (ISI) | 1 week after starting treatment.
  Self-administered questionnaire of 8 items on a Likert scale from 0 (none) to 4 (Very severe), which assesses nighttime symptoms, sleep quality, and daytime symptoms of insomnia; it has a reliability of 0.82 in its original version; and it has similar psychometric indicators in a version validated in Spanish. In its version for the Mexican population, it obtained a 0.84 reliability coefficient.
SF-36 Health Survey | 1 week after starting treatment.
  It is a self-applicable instrument that evaluates the quality of life of people, it is divided into 8 dimensions associated with health such as: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. Each of these dimensions is evaluated in a different way, being a Likert scale between 4 and 5 response options and dichotomous (yes/no) in others. Within the Mexican version, the psychometric properties showed a high internal consistency with a Cronbach's alpha of 0.93.
Generalized Anxiety Disorder 7 (GAD-7) | 1 week after starting treatment.
  Self-administered questionnaire that assesses the presence and severity of generalized anxiety symptoms. It is made up of 7 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range from 0 to 21. It is interpreted that a score greater than 10 is considered as generalized anxiety. Within its psychometric properties, the version translated into Spanish has a high internal consistency with a Cronbach's alpha of 0.8.

SECONDARY OUTCOMES:
Sleep diary | 4 weeks after starting treatment
  Self-registration format subjectively evaluates the number of sleepless nights, subjective sleep quality, number of awakenings per night, sleep onset latency, and sleep efficacy
Patient Health Questionnaire 9 (PHQ-9) | 4 weeks after starting treatment
  Self-applied questionnaire that assesses the presence and severity of depressive symptoms. It is made up of 9 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range of 0 to 27. These scores are interpreted from 0 to 5 (mild), 6 to 10 (moderate), 11 to 15 (moderately severe) and 16 to 27. (severe). Within its psychometric properties, the original version has a high internal consistency with a Cronbach's alpha of 0.86, while the Mexican version was 0.89.
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks after starting treatment
  Self-administered questionnaire that assesses sleep quality. It is made up of 24 reagents; the total score has a range of 0 to 21 points; where a total score less than 5 points indicates good sleep quality and a score greater than 5 points is interpreted as poor sleep quality. In the Mexican population, he obtained a Cronbach's Alpha of 0.78.
Insomnia Severity Index (ISI) | 4 weeks after starting treatment
  Self-administered questionnaire of 8 items on a Likert scale from 0 (none) to 4 (Very severe), which assesses nighttime symptoms, sleep quality, and daytime symptoms of insomnia; it has a reliability of 0.82 in its original version; and it has similar psychometric indicators in a version validated in Spanish. In its version for the Mexican population, it obtained a 0.84 reliability coefficient.
SF-36 Health Survey | 4 weeks after starting treatment
  It is a self-applicable instrument that evaluates the quality of life of people, it is divided into 8 dimensions associated with health such as: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. Each of these dimensions is evaluated in a different way, being a Likert scale between 4 and 5 response options and dichotomous (yes/no) in others. Within the Mexican version, the psychometric properties showed a high internal consistency with a Cronbach's alpha of 0.93.
Generalized Anxiety Disorder 7 (GAD-7) | 4 weeks after starting treatment
  Self-administered questionnaire that assesses the presence and severity of generalized anxiety symptoms. It is made up of 7 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range from 0 to 21. It is interpreted that a score greater than 10 is considered as generalized anxiety. Within its psychometric properties, the version translated into Spanish has a high internal consistency with a Cronbach's alpha of 0.8.
Sleep diary | follow-up 3 months after the end of treatment
  Self-registration format subjectively evaluates the number of sleepless nights, subjective sleep quality, number of awakenings per night, sleep onset latency, and sleep efficacy
Patient Health Questionnaire 9 (PHQ-9) | follow-up 3 months after the end of treatment
  Self-applied questionnaire that assesses the presence and severity of depressive symptoms. It is made up of 9 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range of 0 to 27. These scores are interpreted from 0 to 5 (mild), 6 to 10 (moderate), 11 to 15 (moderately severe) and 16 to 27. (severe). Within its psychometric properties, the original version has a high internal consistency with a Cronbach's alpha of 0.86, while the Mexican version was 0.89.
Pittsburgh Sleep Quality Index (PSQI) | follow-up 3 months after the end of treatment
  Self-administered questionnaire that assesses sleep quality. It is made up of 24 reagents; the total score has a range of 0 to 21 points; where a total score less than 5 points indicates good sleep quality and a score greater than 5 points is interpreted as poor sleep quality. In the Mexican population, he obtained a Cronbach's Alpha of 0.78.
Insomnia Severity Index (ISI) | follow-up 3 months after the end of treatment
  Self-administered questionnaire of 8 items on a Likert scale from 0 (none) to 4 (Very severe), which assesses nighttime symptoms, sleep quality, and daytime symptoms of insomnia; it has a reliability of 0.82 in its original version; and it has similar psychometric indicators in a version validated in Spanish. In its version for the Mexican population, it obtained a 0.84 reliability coefficient.
SF-36 Health Survey | follow-up 3 months after the end of treatment
  It is a self-applicable instrument that evaluates the quality of life of people, it is divided into 8 dimensions associated with health such as: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. Each of these dimensions is evaluated in a different way, being a Likert scale between 4 and 5 response options and dichotomous (yes/no) in others. Within the Mexican version, the psychometric properties showed a high internal consistency with a Cronbach's alpha of 0.93.
Generalized Anxiety Disorder 7 (GAD-7) | follow-up 3 months after the end of treatment
  Self-administered questionnaire that assesses the presence and severity of generalized anxiety symptoms. It is made up of 7 items on a Likert scale that goes from 0 (not at all) to 3 (almost every day). The evaluation consists of the sum of the scores of each item having a range from 0 to 21. It is interpreted that a score greater than 10 is considered as generalized anxiety. Within its psychometric properties, the version translated into Spanish has a high internal consistency with a Cronbach's alpha of 0.8.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio B Álvarez García, M.D, Principal Investigator — Sleep Disorder Clinic
Locations (1):
- Horacio Balam Álvarez García, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The database will be kept by the researchers and will be shared with other researchers upon request.

REFERENCES:
- [Result] Ahmad SJ, Feigen CM, Vazquez JP, Kobets AJ, Altschul DJ. Neurological Sequelae of COVID-19. J Integr Neurosci. 2022 Apr 6;21(3):77. doi: 10.31083/j.jin2103077. PMID 35633158
- See also: Neurological Sequelae of COVID-19 — https://www.imrpress.com/journal/JIN/21/3/10.31083/j.jin2103077